CLINICAL TRIAL: NCT00168259
Title: Evaluation of Interferon-gamma Responses to HCMV Infection in HIV Positive Individuals
Status: Completed | Type: Observational
Sponsor: The Alfred (Other)
Collaborators: Cellestis (Industry)
Responsible Party: Principal Investigator, Jennifer Hoy, Professor Jennifer Hoy, The Alfred
Other Study IDs: 185/04
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: HIV Infection; CMV Infection
Keywords: Treatment Naive; HIV
MeSH Terms: conditions — HIV Infections; Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, and DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
The study is designed to evaluate interferon responses to CMV in HIV positive individuals and a component will look at interferon responses to CMV in HIV positive individuals over time after commencement of antiretroviral therapy. We will also look at the correlation between CD4 T cell numbers and HLA type with the interferon response.

ELIGIBILITY:
Inclusion Criteria:

1. HIV positive with history of documented HCV infection
2. Over 18 years old
3. HIV positive
4. Antiretroviral naive, starting on antiretroviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV infected patients with past CMV infection initiating antiretroviral therapy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2004-12; Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Lewin, Professor, Principal Investigator — The Alfred
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia